CLINICAL TRIAL: NCT05394246
Title: Intraoperative Liver Tumor Imaging Using Fluorescent-labeled Human IgG
Brief Title: Fluorescent-labeled IgG for Liver Tumor Detection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Sciences (Other Government)
Responsible Party: Principal Investigator, Zeyu Zhang, PHD, Principal Investigator, Chinese Academy of Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FluoAB-Liver
Record Dates: First submitted 2022-05-19; First posted 2022-05-27 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FluoAB intraoperative fluorescence imaging (Experimental): The patients will receive an injection of FluoAB. Surgery will be performed with guidance by FluoAB fluorescence imaging.
  Interventions: Drug: FluoAB

INTERVENTIONS:
Drug: FluoAB — Drug Injection: FluoAB (fluorescent-labeled IgG)

SUMMARY:
This study is to evaluate whether intraoperative fluorescence imaging using fluorescent-labeled IgG probe (FluoAB) can help distinguish the tumor and the liver cirrhosis (or the liver parenchyma).

The main purposes of this study include:

* To validate the safety and effectiveness of using FluoAB in hepatic surgery.
* To raise the surgical precision with guidance by FluoAB fluorescence imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been diagnosed with liver tumor.
2. Planned to receive hepatectomy.
3. Liver function Child-Pugh A/B.
4. The expected lifetime is longer than 6 months.
5. Approved to sign the informed consent.

Exclusion Criteria:

1. Enrolled in other trials in the past 3 months.
2. Metastatic lesions were found.
3. Undesirable function of heart, lung, kidney, or any other organs.
4. Unable to tolerate a hepatectomy.
5. The researchers considered inappropriate to be included.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Tumor imaging precision | Update with an average of 2 weeks.
  Sensitivity and specificity of hepatic malignancy detection by fluoAB intraoperative imaging.
Tumor lesions | Immediately after the hepatic surgery.
  Numbers of intraoperatively detected tumor lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Li, MD., Principal Investigator — The Affiliated Hospital Of Southwest Medical University
Locations (1):
- The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan, China